CLINICAL TRIAL: NCT02297113
Title: The C-MAC Videolaryngoscope Compared With Conventional Laryngoscopy for Rapid Sequence Intubation at the Emergency Department
Brief Title: Rapid Sequence Intubation at the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEK Zurich 2014-0356
Record Dates: First submitted 2014-11-13; First posted 2014-11-21 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Emergency
Keywords: patients; departement; requiring Rapid Sequence Intubation (RSI)
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional endotracheal intubation (Active Comparator): Patients assigned to this group will be intubated using conventional Macintosh blade in adequate size.
  Interventions: Device: Macintosh blade
- C-MAC (Active Comparator): Patients assigned to this group will be intubated using C-MAC videolaryngoscope in adequate size.
  Interventions: Device: C-MAC videolaryngoscope

INTERVENTIONS:
Device: Macintosh blade — conventional endotracheal intubation
  Arms: conventional endotracheal intubation
Device: C-MAC videolaryngoscope
  Arms: C-MAC

SUMMARY:
All patients undergoing emergent endotracheal intubation (RSI) at the Emergency Department will be screened for inclusion in this clinical study. The indication of endotracheal intubation is an exclusively clinical decision and is not affected by this study protocol in any aspect.

If fulfilling the In- and exclusion criteria's, patient will be randomly assigned to one of two groups

1. C-MAC Videolaryngoscope in appropriate size
2. conventional endotracheal intubation using Macintosh Blade in appropriate size

Randomization (1:1) will be based on computer-generated codes maintained in sequentially numbered opaque envelopes that will be opened immediately before randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring emergency Rapid Sequence Intubation at the emergency department
* Male and Female subjects 18 years to 99 years of age
* Written confirmation by a physician not involved in this study
* Written informed consent by the participant (obtained afterwards)
* Patient not showing remarkable rejection in participation in this study

Exclusion Criteria:

* Maxilla-Facial trauma
* Immobilized cervical spine
* Indication for fiberoptic guided intubation (known difficult airway)
* Ongoing Cardio-Pulmonary-Resuscitation (CPR)
* Involvement in any other clinical trial during the course of this trial, within a period of 30 days prior to its beginning or 30 days after its completion
* Severe or immediately life-treating injury requiring immediate medical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Success Rate | 10 minutes
  defined as successful placement of endotracheal tube within the trachea and

SECONDARY OUTCOMES:
time to intubation | 10 minutes
  defined as time between insertion of the videolaryngoscope/ Macintosh blade into the mouth until detection of end-tidal CO2
Laryngoscopic view | 10 minutes
  Cormack and Lehane Score
Number of intubation attempts | 10 minutes
Unrecognized esophageal intubation | 10 minutes
Ease of intubation (1-5) | 10 minutes
  o (1) very easy, (2) easy, (3) somewhat difficult, (4) difficult, (5) impossible
Violations of the teeth | 10 minutes
  number of patients; teeth will be inspected for potential damage and documented accordingly
Necessity of using further, alternative airway devices for successful intubation (if randomized airway device failed) | 10 minutes
  number of patients, requiring alternate device
Maximum drop of saturation | 10 minutes
  Spo2 will be measured continuously and documented accordingly

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zuerich, Dept of Anesthesiology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Sulser S, Ubmann D, Brueesch M, Goliasch G, Seifert B, Spahn DR, Ruetzler K. The C-MAC videolaryngoscope compared with conventional laryngoscopy for rapid sequence intubation at the emergency department: study protocol. Scand J Trauma Resusc Emerg Med. 2015 Apr 24;23:38. doi: 10.1186/s13049-015-0119-x. PMID 25903358
- [Derived] Sulser S, Ubmann D, Schlaepfer M, Brueesch M, Goliasch G, Seifert B, Spahn DR, Ruetzler K. C-MAC videolaryngoscope compared with direct laryngoscopy for rapid sequence intubation in an emergency department: A randomised clinical trial. Eur J Anaesthesiol. 2016 Dec;33(12):943-948. doi: 10.1097/EJA.0000000000000525. PMID 27533711